CLINICAL TRIAL: NCT04813497
Title: Monitoring of COVID-19 Seroprevalence Among GHdC Staff Members: Protocol for an Interventional Cohort Study in 2020-2021
Brief Title: Monitoring of COVID-19 Seroprevalence Among GHdC Staff Members
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Grand Hôpital de Charleroi (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: SARS-COV-2-SERO_FU-2021_GHdC
Record Dates: First submitted 2021-03-21; First posted 2021-03-24 (Actual); Last update posted 2022-06-01 (Actual); Status verified 2022-05

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Intervention Model Description: Group 1 : participants who did not agree to receive a SARS-CoV-2 vaccine in the first Belgian campaing but who agreed to perform a serological test against COVID-19.
  Groups of participants who agree to receive a SARS-CoV-2 vaccine at different specific times determined by the Belgian State for workers at the Grand Hôpital de Charleroi.
  Parallel study of immunity to SARS-CoV-2 among staff members.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Participants who refuse the SARS-CoV-2 vaccine (Other): Participant who does not wish to be vaccinated against the SARS-CoV-2 virus and who wishes to perform the serological test during the vaccination campaign and the second 12-14 weeks after the first serological test.
  Interventions: Diagnostic Test: Serology to determine SARS-CoV-2 infection
- Participants who received the first dose of SARS-CoV-2 vaccine before the first serological test (Other): Participant who has received his first dose of vaccine and who performs his serological test when he receives the second dose of vaccine against the SARS-CoV-2 virus to determine his immunity. The second serological test will be done 12 to 14 weeks after the second dose of the SARS-CoV-2 vaccine to determine its immunity.
  Interventions: Diagnostic Test: Serology to determine SARS-CoV-2 infection
- Participants who start with the serological test before SARS-CoV-2 vaccine (Other): Participant who performed the serological test before the first dose of vaccine and 12 to 14 weeks after the second dose of vaccine against the SARS-CoV-2 virus to determine his immunity.
  Interventions: Diagnostic Test: Serology to determine SARS-CoV-2 infection
- Participants who received the third dose of SARS-CoV-2 vaccine (Other): Participant who performs his serological test when he receives the third dose of vaccine against the SARS-CoV-2 virus to determine his immunity.
  Interventions: Diagnostic Test: Serology to determine SARS-CoV-2 infection
- Participant who received the third dose of SARS-CoV-2 vaccine and (Other): Participant who performs a serological test between 12 and 14 weeks after the third dose of SARS-CoV-2 vaccine to determine immunity. And who has agreed to undergo serological testing prior to the third dose of the vaccine.
  Interventions: Diagnostic Test: Serology to determine SARS-CoV-2 infection

INTERVENTIONS:
Diagnostic Test: Serology to determine SARS-CoV-2 infection — Each participant accept to have two blood tests on a dry tube of maximum 8 ml of whole blood

SUMMARY:
Grand Hôpital de Charleroi (GHdC) had to organize the vaccination of its staff in December 2021 against SARS-CoV-2.On the sidelines of this vaccination campaign, the management committee agreed to document the knowledge of the SARS-CoV-2 serology of all the staff of the establishment before this vaccination campaign, as well as a few weeks after vaccination.

In November 2021, the Belgian government decided to offer a third dose of vaccine against SARS-CoV-2 virus. The GHdC managment committee has agreed to continue monitoring SARS-CoV-2 serology for members who receive their third dose of vaccine.

DETAILED DESCRIPTION:
Grand Hôpital de Charleroi (GHdC) staff were exposed to the risk of SARS-CoV-2 infection during the first half of 2020: a seroprevalence survey, conducted in the summer of 2020, after the "first wave" of the epidemic, and before the "second wave", thus revealed a significant seroprevalence because of its exposure. This study, because of its high participation rate, also showed the sustained interest of the agents in knowing their serology, either for personal reasons, or for the purposes of recognition as an occupational disease.

The GHdC decided in December 2020 to organize as soon as possible the vaccination of its salaried and self-employed employees who wish to take advantage of this opportunity. On the sidelines of this vaccination campaign, the management committee agreed to document the knowledge of the SARS-Cov-2 serology of all the staff of the establishment before this vaccination campaign, as well as a few weeks after vaccination. This knowledge must better organize the disease prevention strategy, both with regard to the staff themselves and the patients for whom they are called upon to treat.

When the Belgian government decided in November 2021 to offer a third dose of vaccine and start it up in hospitals, the GHdC managment committee has agreed to continue monitoring SARS-CoV-2 serology for members who agree to receive their third dose of vaccine.

ELIGIBILITY:
Inclusion Criteria:

* To be an employee or independent collaborator at the GHdC

Exclusion Criteria:

* Refusal to take a blood test for anti-SARS-CoV-2 antibodies

Regarding amendment 1:

* Members who did not receive the third dose of PFIZER vaccine (Comirnaty) during the GHdC vaccination campaign and who did not performed a blood test to measure anti-SARS-CoV-2 antibodies.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 4000 (Actual)
Dates: Start 2021-02-05 (Actual); Primary Completion 2022-04-30 (Actual); Study Completion 2022-04-30 (Actual)

PRIMARY OUTCOMES:
Serological tests to know the level of antibodies against SARS CoV-2 | up to 14 weeks after the second dose of SARS-CoV-2 vaccine or after the first serological test
  Participants accept to undergo 2 serological tests to determine their immunity to the SARS-CoV-2 virus.

CONTACTS AND LOCATIONS:
Overall Officials: Natahie de Visscher, MD, Principal Investigator — Grand Hôpital de Charleroi
Locations (1):
- Grand Hôpital de Charleroi, Charleroi, Hainaut, Belgium

IPD SHARING:
Plan to Share IPD: No